CLINICAL TRIAL: NCT01325727
Title: Brief Computerized Feedback for Smokers in Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HM13510
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Smoking
MeSH Terms: conditions — Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief computerized feedback (Experimental): Brief computerized feedback
  Interventions: Other: Brief computerized feedback
- Resources only (Active Comparator)
  Interventions: Other: Resources only (control)

INTERVENTIONS:
Other: Brief computerized feedback — Brief computerized feedback
  Arms: Brief computerized feedback
Other: Resources only (control) — Participants randomized to the control group will discuss the option of quitting smoking, along with an information sheet, highlighting resources available to assist participants with smoking cessation, such as the Virginia Quitline (1-800 QUIT NOW) and nicotine replacement therapy.
  Arms: Resources only

SUMMARY:
The purpose of this research study is to find out more about smokers in recovery from addiction to alcohol/other drugs, and to evaluate a brief computerized smoking behavior feedback session. The hypothesis is that a brief computerized smoking behavior feedback session will motivate more smokers to quit smoking than a control condition.

ELIGIBILITY:
Inclusion Criteria:

1. Be 18 years of age or older
2. Be in recovery from addiction to alcohol and/or drugs (self-defined)
3. Have smoked at least one cigarette per day for the past seven days or at least 10 cigarettes total during the past week
4. Have smoked at least 100 cigarettes (lifetime)
5. Have an expired air carbon monoxide (CO) level of > 6 ppm (verifies current smoking)
6. Be cognitively able to understand the proposed research design (screening followed by random assignment to one of the two conditions, if appropriate)

To be eligible to receive NRT (if chosen by the participant), participants must:

1. Not be pregnant, breastfeeding, or plan to become pregnant in the next year
2. Not have experienced a myocardial infarction (heart attack) or have been hospitalized for a heart-related problem in the last 2 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
% quit smoking | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alison Breland, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Substance Abuse Addiction and Recovery Alliance Center, Midlothian, Virginia, United States